CLINICAL TRIAL: NCT05812560
Title: Evaluation of a Protocolposturalchanges in Women Giving Birth Whith Epidural Analgesia. Clinical Trial.
Brief Title: Evaluation of a Protocol Posturalchanges in Women Giving Birth With Epidural Analgesia. Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, María de la Milagrosa Fontan Azpeitia, University degree in nursing specializing in obstetrics and gynecology, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PI 176/21
Record Dates: First submitted 2023-02-10; First posted 2023-04-13 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Epidural Analgesia; Nulliparous Pregnant; Labor With Postural Changes; Randomized
Keywords: Movement; Postural change; Childbirth; Epidural analgesia.

STUDY DESIGN:
Intervention Model Description: Pregnant women will make 2 postural changes every 60 min throughout labor, preferably every 30 min.
  The positions will be different depending on the phase of labor in which the pregnant woman is. Those that correspond to each period have been chosen based on the comfort of the woman. These positions are set out below, finding in annex 3 more details of them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervetion (Experimental): The intervention of the experimental group: application of a protocol of postural changes every 30-60 min or at least two postural changes in one hour during labor.
  Interventions: Other: postural changes
- Control (No Intervention): In the control group, each midwife will apply postural changes according to their usual practice. Differences with the experimental group: the choice of postural changes according to the stage of labor, its cadence and posture during the expulsive.

INTERVENTIONS:
Other: postural changes — application of a protocol of postural changes every 30-60 min or at least two postural changes in one hour during labor.
  Arms: Intervetion

SUMMARY:
. The pain that occurs during labor is controlled in our environment through epidural analgesia.

This mainly generates a sensory block but also a motor block that suppresses different reflexes physiological factors that facilitate the development of childbirth.

Being necessary to adapt obstetric care to this reality. Among which are the changes postures of the immobile pregnant woman. General Objective: To evaluate the impact of a mobilization protocol during labor in pregnant women with epidural analgesia versus usual mobilization.

Material and method Simple randomized clinical trial, in a 1:1 ratio. Population: nulliparous pregnant women and low-risk pregnancy, using epidural analgesia.

Inclusion criteria: nulliparous pregnant women at term and low-risk pregnancy, in the active phase of labor and with epidural analgesia, voluntarily participating in the study.

Sample size: Assuming an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided contrast, each group will contain 104 subjects to detect a difference 0.4 units.

The intervention of the experimental group will consist of the application of a protocol of postural changes every 30-60 minutes or at least two postural changes in one hour during labor, in order to expand the diameters pelvics in the different phases of this.

In the control group, each midwife will apply the postural changes according to her usual practice.

Differences with the experimental group: the choice of postural changes according to the stage of labor, its cadence and the posture during the expulsive.

DETAILED DESCRIPTION:
Justification:

Variability in clinical practice in this setting ranges from no postural changes at all, random postural changes unrelated to stage of labor, to changes frequently targeted at each stage of labor, with knowledge of the pelvis and the mechanisms of childbirth.

There are no validated procedures for mobilizing pregnant women with epidural analgesia during labor. This makes investigators think about the need to design a protocol for postural changes during labor and the training of the team of midwives. All of this aimed at offering unified and quality care to pregnant women, which is not only reversed in maternal-fetal results but also in greater maternal comfort and in the perception of quality care by the pregnant woman.

In this study we will focus on mitigating the motor effects of epidural analgesia on labor and expulsive periods by establishing standardized postural changes.

Hypothesis and objectives:

The implementation of a protocol that standardizes postural changes during labor in nulliparous pregnant women with epidural analgesia will have an impact on dilation and expulsive times, improving obstetric and perinatal outcomes that are universally measured with the type of delivery, the perineal status, the apgar test at one minute and ten minutes of neonatal life and the ph result of umbilical cord blood. 9 General objective to evaluate the impact of a mobilization protocol during labor versus conventional mobilization in nulliparous pregnant women with epidural analgesia.

Specific objectives

* Evaluate the speed of dilation and expulsive time in both situations.
* Record the need for artificial amniorrhexis and oxytocin perfusion in both situations.
* Analyze the type of delivery according to the group to which the pregnant woman belongs.
* Examine the perineal state after childbirth in both situations.
* Evaluate the behavior of variables related to the extrauterine adaptation of the newborn in both groups: apgar test, neonatal resuscitation, ph in blood from the umbilical artery or vein.

Methodology:

type of study Simple randomized clinical trial with parallel groups, single center, carried out in a tertiary hospital of the Madrid Health Service. Participants will be randomly assigned to each of the groups in a 1:1 ratio. Randomization will be carried out using a list of random numbers with the Epidad program (version 3.1) and masking using sealed and sequentially numbered envelopes.

Study population Nulliparous pregnant women with a low risk in the evolution of the gestation17 who make use of epidural analgesia and go to the hospital under study for delivery care.

Inclusion, exclusion and elimination criteria Pregnant women older than 18 years, nulliparous at term and low risk in pregnancy will be included17. They must be in the active phase of labor (3 cm dilated and regular contractions every 2-3 minutes9), with the intention of using epidural analgesia, showing no contraindications for such anesthesia, and wishing to participate voluntarily in the study.

Those pregnant women who, during labor, the midwife cannot complete the registration, due to workload or the woman decides to abandon participation in the study, will be excluded.

Those participants in the experimental group who, for obstetric, maternal or fetal comfort reasons, cannot follow the protocol for postural changes will be eliminated from the study.

Sample size Accepting an alpha risk of 0.05 and a beta risk of 0.2 on a two-sided contrast, it takes 104 subjects in each arm to detect a difference of 0.4 time units. The common standard deviation is assumed to be 1. A rate of loss to follow-up of 5% has been estimated. Data extrapolated from previous studies. 19 (calculated using the program grammo V.7.12) Main Variable • Time of labor: the time in minutes that elapses of labor will be recorded (dilation phase + expulsive phase). For this, a bodet brand digital clock will be used, which will be calibrated every 24 hours. The dilation phase will be measured as dilation velocity in cm/h and the expulsive phase in min.

1. Dilation time: period of labor that elapses between 4 and 10 cm of dilation and is accompanied by regular dynamics.
2. Expulsive time in minutes: period of labor that elapses between the moment in which full dilation is reached (10 cm of cervical dilation) and the moment in which fetal expulsion occurs.

Secondary Variables

* Cervical dilation: opening of the uterine cervical opening. It will be measured through vaginal examination and the unit will be centimeters, it will be recorded every two hours throughout the labor in both groups.
* Type of amniorhexis: rupture of the amniotic bag, it can be of two types:

artificial (when carried out by the midwife or obstetrician using a sterile amniorhexis lancet): if cervical dilation in 4 hours < 2 cm with amniotic bag integrates, perform artificial amniorrhexis and if after two hours cervical dilation is < 1 cm administer oxytocin910 spontaneous: In this case, a dose of oxytocin will be administered according to the international recommendation of clinical practice guidelines10.

It will be recorded only once when it happens.

* Use of oxytocin: the use or not of oxytocin at the end of labor will be recorded, as well as the amount in IU/kg/hour administered,
* Type of delivery: eutocic delivery, which is one that does not require medical intervention.

Dystocic delivery, after a change in normality, requires an obstetric intervention, which may be: instrumental (if an obstetric instrument such as forceps, spatulas, or a suction cup is used to extract the fetus) or caesarean section (when a consistent surgical intervention is carried out). in fetal extraction through an incision in the abdomen of the pregnant woman to access the uterine cavity). It will be recorded at the end of delivery.

* Umbilical cord blood pH: analysis of umbilical cord blood is an objective measure of fetal condition before birth. The spanish association of pediatrics defines serious neurological sequelae in children with arterial pH greater than 720 as infrequent. It will be measured with a rediomether® brand abl90 flex pachymeter (The analyzer incorporates an automatic quality control with specific QC solutions and performs also continuous analytical checks of the system and undertakes automated corrective actions when necessary.). The unit will be numbers with two decimal places and will be recorded at the end of delivery.
* Score in the neonatal apgar test: Evaluates the newborn's adaptation to extrauterine life, scores 5 parameters in the newborn: heart rate, respiratory effort, muscle tone, response to stimuli and skin color. Each parameter is given a score of 0.1 or 2. The maximum score will be 10 and the minimum 0. An apgar test above 7 indicates a good adaptation to extrauterine life. An integer number from 0 to 10 will be recorded, at one minute and at 5 minutes of the neonate's life. twenty-one
* Need for neonatal resuscitation and type: It is related to the need to apply support measures to the newborn for its adaptation to extrauterine life. It will be measured in numbers with a decimal from 0 to 5 according to the application of no measure 0, aspiration of airway secretions 1, application of continuous positive airway pressure 2, application of intermittent positive airway pressure 3, application of orotracheal intubation 4, drug administration 5. It will be recorded according to the type after 10 minutes of the newborn's life. twenty-one.

Personal variables

* Age: it will be measured in years
* Obstetric history: pregnancies, abortions, deliveries and living children. It will be measured in whole numbers.

Gestational age: time that elapsed from the date of the last period of the pregnant woman until her recruitment for the study, will be measured in whole weeks.

Recruitment and management of pregnant women

1. The recruitment of the pregnant woman will be carried out upon admission to the delivery unit by the responsible collaborating midwife.
2. The pregnant woman will be given the information sheet (annex 4) and two copies of the informed consent (annex 5).
3. Once the pregnant woman carefully reads the study information and resolves her doubts with said midwife, she will collect one of the signed copies of the informed consent, the other will belong to the pregnant woman.
4. When participant proceed to grant his written consent, participant will be randomly assigned to belong to the control group or the intervention group at random. The randomization process will be carried out by all the women who come to our center and agree to participate in the study, with prior information (annex 4) and sign the informed consent (annex 5). Once recruited, the participants will have a number, avoiding revealing the participant's personal data. Through the data collection notebook, the number assigned to the study subject, the obstetric data of the pregnant woman and the variables described above will be recorded.

Preparation Preparation of the midwives: the midwives who are part of the study must have a minimum of 10 years' experience in assisting women in childbirth, as well as training in obstetric simulation. They will be informed of the object of the study (annex 1) and will receive training to standardize data collection. The total number of midwives will be divided into two groups: 1. Those who will carry out mobilizations according to their usual practice and 2. Those who will carry out the experimental mobilization protocol, which will receive a specific training module to be able to carry it out.

Training for professionals: to standardize data collection, training will be provided to all professionals participating in the study. This training will consist of 3 sections:

1. Introduction; 2. Necessity and justification of the investigation; 3. Practical examples for training in the collection of variables (Annex 2).

   The session will be held online and its duration will be one hour. The midwives of the experimental group, in addition to general training, will receive a separate face-to-face module to be able to carry out the experimental mobilization protocol. In this session, the different positions will be explained and training will be carried out through simulated cases. The session will last 2 hours.

   Intervention experimental group. Mobilization protocol: Pregnant women will make 2 postural changes every 60 min throughout labor, preferably every 30 min.

   The positions will be different depending on the phase of labor in which the pregnant woman is. Those that correspond to each period must be chosen based on the comfort of the woman. These positions are set out below, finding in annex 3 more details of them.

   A) Active phase of dilation (vaginal examination >4 cm and <10 cm). The following positions must be adopted:
   * sims
   * Sitting with knee external rotation
   * Walchers
   * Modified lateral prone

   B) Passive expulsive phase (vaginal examination ≥10 cm without contractions). The following positions must be adopted:

   -sims
   * Sitting with knee external rotation
   * Walchers
   * Modified lateral prone
   * modified sims
   * Sitting with knee internal rotation
   * Lateral decubitus with knee external rotation
   * On knees with parallel or symmetrical legs
   * McRoberts semi-sitting.

   C) Active expulsive phases (vaginal examination ≥10 cm with contractions). The following positions must be adopted:

   - modified sims

   - Sitting with knee internal rotation
   * Lateral decubitus with knee external rotation
   * On knees with parallel or symmetrical legs
   * McRoberts semi-sitting. Control group: the midwife will develop postural changes according to her usual practice. The existence of postural changes or not and the time spent in each of the chosen positions will be recorded.

   In both groups, from the beginning of labor until the end of it, the midwife will perform a vaginal examination every 2 hours, evaluating the stage of labor in which the pregnant woman is.

   Once the delivery is over, the responsible midwife will file the informed consent and the data notebook.

   Ethical aspects The study will be carried out in accordance with the declaration of Helsinki, compliance with the biomedical research law and compliance with good clinical practice standards, which include study monitoring to ensure data quality and subject protection. participants. The study protocol will be reviewed and approved by the huphm clinical research ethics committee. Before beginning any procedure, the informed consent of the participants will be obtained. The confidentiality of the information and the anonymity of the participants will be guaranteed in compliance with organic law 3/2018, of december 5, on the protection of personal data and guarantee of digital rights.

   Limitations and strengths of the study Limitations: double blinding. The complete application of the protocol due to the influence of foreign variables such as: maternal or fetal comfort or the type of delivery such as an instrumental delivery.

   The variability in the assessment of cervical dilation, which was attempted to be alleviated with the experience and simulation training of midwives.

   Strengths:

   It is a non-bloody intervention, since it is based on the adoption of positions, without having to invade the body or administer poisons for therapeutic purposes.

   If we obtain the desired results, and really as the literature suggests, this intervention contributes to improving obstetric and perinatal outcomes, it will have a great impact on the quality of care offered to pregnant women and their children. And it can be quickly implemented by the entire obstetric team given the simplicity of the postural change protocol.

   Means available to carry out the project • Human resources: nurses specialized in obstetrics and gynecology who wish to participate, belonging to the obstetric block team at huph Majadahonda.

   • Material means: necessary stationery for data collection notebooks, information sheets, protocol.

   Study development schedule • Documentary support and CEIC. Duration 7 months Administrative procedures: review of the data collection Notebook (CRD) and the mobilization protocol by the midwives of the research team.

   Presentation of the study to the clinical research ethics committee of the puerta de hierro majadahonda university hospital.

   Pilot Study: a pilot study will be carried out, recruiting 6 pregnant women per group, to evaluate the recruitment procedures, information (hip and ic), randomization, follow-up, completion of the data collection Notebook and information collection. The entire research team will participate in this first stage.

   Communication to the team: in this phase the meeting of researchers will be held, in which the research protocol will be reviewed and the results of the pilot study will be communicated.

   • Patient recruitment and data collection. Duration 12 months depending on the pregnant women who meet the inclusion criteria and the recruitment capacity of the research team. It will be carried out by the midwives who wish to participate in the study, by the midwives of the research team.

   The study will be carried out in the obstetrics service of the puerta de hierro Majadahonda university hospital (Madrid).
   * Review database, sanitation and complete information. Duration 1 months. Simultaneously to the development of stage 2, the quality of the data obtained will be assessed, to complete the missing information and to be able to carry out intermediate analyses.
   * Full analysis, dissemination of results and final report. Duration 2 months Once the 208 study subjects have been recruited, a complete analysis of the database will be carried out for the elaboration of the pertinent manuscripts and the elaboration of the Final Report.

   Once the results of the study are known, the priority is to make them known to the entire Obstetrics Service by presenting them in a Clinical session and delivering an abbreviated report.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women older than 18 years, nulliparous at term and low risk in pregnancy will be included17. They must be in the active phase of labor (3 cm dilated and regular contractions every 2-3 minutes9), with the intention of using epidural analgesia, showing no contraindications for such anesthesia, and wishing to participate voluntarily in the study.

Exclusion criteria:

* Those pregnant women who, during labor, the midwife cannot complete the registration, due to workload or the woman decides to abandon participation in the study, will be excluded.

Those participants in the experimental group who, for obstetric, maternal or fetal comfort reasons, cannot follow the protocol for postural changes will be eliminated from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Cervical dilation speed | From the beginning to the end of the labor 12-24 hours
  The dilation phase will be measured as dilation speed in cm/h,Dilation time: period of labor that elapses between 4 and 10 cm of dilation and is accompanied by regular dynamics
Expulsive time | From the beginning to the end of the labor 12-24 hours
  Expulsive time in minutes: period of labor that elapses between the moment in which full dilation is reached (10 cm of cervical dilation) and the moment in which fetal expulsion occurs.

SECONDARY OUTCOMES:
Type of the delivery | It will be recorded at the end of delivery. 12-24 hours
  Type of delivery: Eutocic delivery, which is one that does not require medical intervention Dystocic delivery, after a change in normality, requires an obstetric intervention, which may be: instrumental (if an obstetric instrument such as forceps, spatulas, or a suction cup is used to extract the fetus) or caesarean section (when a consistent surgical intervention is carried out). in fetal extraction through an incision in the abdomen of the pregnant woman to access the uterine cavity).

CONTACTS AND LOCATIONS:
Locations (1):
- Maria de la Milagrosa Fontan Azpeitia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No